CLINICAL TRIAL: NCT06212492
Title: Effects on Biotrauma of Combining Routine CURArization With Prone Positioning During Adult Acute Respiratory Distress Syndrome
Brief Title: Effects on Biotrauma of NMBAs and PP Association During ARDS
Acronym: CURA-PRONE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCAPHM21_0414; ID-RCB (Other: 2023-A01797-38)
Record Dates: First submitted 2023-12-11; First posted 2024-01-19 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2023-12

CONDITIONS: Moderate to Severe Acute Respiratory Distress Syndrome
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone Positioning and NMBAs (PP-NMBAs) (Experimental): Early and systematic use of Prone positioning and NMBAs
  Interventions: Drug: NMBAs; Other: Prone positioning
- Prone Positioning (PP) (Active Comparator): Early and systematic use of prone positioning with NMBAs indicated ONLY as rescue
  Interventions: Other: Prone positioning

INTERVENTIONS:
Drug: NMBAs — Early and systematic use of NMBAs
  Arms: Prone Positioning and NMBAs (PP-NMBAs)
Other: Prone positioning — Early and systematic use of prone positioning

SUMMARY:
The improved survival of patients with acute respiratory distress syndrome (ARDS) over the last decades is related to the use of so-called "protective" mechanical ventilation. Two therapies have been shown to increase survival among the most hypoxemic patients (PaO2/FiO2 < 150 mmHg): a continuous use of neuromuscular blocking agents (NMBAs) for 48 hours in the acute phase of ARDS and prone positioning (PP). NMBAs and PP are part of the latest guidelines from French ICU Society. However, North American guidelines recommend PP for patients with severe ARDS only but not NMBAs, given the results of the ROSE study which did not confirm the benefit on mortality demonstrated in the ACURASYS study. However, in the ROSE study, ventilatory strategy, use of NMBAs and PP were different from the ACURASYS study.

Yet, NMBAs and PP are frequently associated in clinical practice, particularly with the COVID-19 pandemic, but also in randomized trials. In the PROSEVA study, almost all the patients (91%) received a continuous infusion of NMBAs during PP. Indeed, there is a common physiopathological rationale in both techniques: they favor the homogenization of transpulmonary pressures (TPP), reduce lung overdistension, Pendelluft effect and thus ventilator induced lung injury (VILI), in particular barotrauma and biotrauma. This reduction of biotrauma has been demonstrated for PP and NMBAs separately, but never by comparing the combined effect of the 2 techniques to each of them separately. This comparison requires reliable tools. In recent years, the "soluble form of the receptor for advanced glycation end products" (sRAGE), a new biomarker specific of pulmonary epithelial aggression and therefore of biotrauma, has been described and evaluated during ARDS and appears to be associated with the severity of pulmonary damage and prognosis.

Overall, despite an interesting physiopathological rationale and a clinically widespread practice, there is currently no study evaluating the synergistic effect of PP and NMBAs in the treatment of ARDS, in particular on the prevention of VILI, and more precisely of biotrauma. This question seems crucial to better specify the respective place of each of these treatments in the management strategy of ARDS patients whose prevalence and mortality remain high.

The objective of this study is therefore to evaluate, using a recent and reliable biomarker, the synergistic effect of a short-term NMBAs infusion using cisatracurium and PP on the reduction of biotrauma during moderate to severe ARDS. The investigators will compare this "synergistic" treatment to the use of PP alone. They will also evaluate, in secondary objectives, the effects of PP and NMBAs combination on clinical outcomes and on the patients' prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Written informed consent of proxy to the study participation
* Invasive mechanical ventilation for ≤ 72 hours at inclusion
* Criteria of moderate to severe ARDS according to the Berlin definition
* Patients covered by or having the rights to social security

Exclusion Criteria:

* Pregnant or breast-feeding women, patients deprived of freedom or under legal authority
* Patients having undergone previous PP sessions during the same stay
* Patients who had already been curarized prior to inclusion
* Patient currently receiving ECMO or any technique of extracorporeal CO2 removal at the time of inclusion
* Patient with a contraindication to PP
* Previous hypersensitivity or anaphylactic reaction to any NMBA
* Chronic respiratory insufficiency with oxygen or long-term ventilation
* SAPS II score at the time of enrollment > 75
* Patients who are moribund or for whom limitations of active therapies have been decided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Difference between the plasma sRAGE value at the end of the first PP session and the baseline value before PP (∆ sRAGE). | Day 1
  Our primary outcome will be the comparison of the differences in plasma sRAGE levels before and after the first PP session (∆ sRAGE), a kinetic being probably more relevant than a raw value, given the observed inter-individual variations of sRAGE at basal state.

SECONDARY OUTCOMES:
Plasma determination of IL1 before the first PP session | Day 1
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of IL1 1 hour after PP initiation at the first PP session | Day 1
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of IL1 at the end of the first PP session | Day 1
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of IL1 4 hours after return to supine after the first PP session | Day 2
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of TNFα before the first PP session | Day 1
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of TNFα 1 hour after PP initiation at the first PP session | Day 1
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of TNFα at the end of the first PP session | Day 1
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of TNFα 4 hours after return to supine after the first PP session | Day 2
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of sRAGE before the first PP session | Day 1
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of sRAGE 1 hour after PP initiation at the first PP session | Day 1
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of sRAGE at the end of the first PP session | Day 1
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of sRAGE 4 hours after return to supine after the first PP session | Day 2
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of angiopoietin 2 before the first PP session | Day 1
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of angiopoietin 2 1 hour after PP initiation at the first PP session | Day 1
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of angiopoietin 2 at the end of the first PP session | Day 1
  Inflammation, pulmonary epithelial and endothelial dysfunction
Plasma determination of angiopoietin 2 4 hours after return to supine after the first PP session | Day 2
  Inflammation, pulmonary epithelial and endothelial dysfunction
PaO2/FiO2 before each PP session | Up to Day 28
  Hematosis
PaO2/FiO2 1 hour after PP initiation at each PP session | Up to Day 28
  Hematosis
PaO2/FiO2 6 hours after PP initiation at each PP session | Up to Day 28
  Hematosis
PaO2/FiO2 at the end of each PP session | Up to Day 28
  Hematosis
PaO2/FiO2 4 hours after return to supine after each PP session | Up to Day 28
  Hematosis
PaO2/FiO2 48 hours after inclusion | 48 hours after inclusion
  Hematosis
PaO2/FiO2 72 hours after inclusion | 72 hours after inclusion
  Hematosis
PaO2/FiO2 7 days after inclusion | 7 days after inclusion
  Hematosis
pH before each PP session | Up to Day 28
  Hematosis
pH 1 hour after PP initiation at each PP session | Up to Day 28
  Hematosis
pH 6 hours after PP initiation at each PP session | Up to Day 28
  Hematosis
pH at the end of each PP session | Up to Day 28
  Hematosis
pH 4 hours after return to supine after each PP session | Up to Day 28
  Hematosis
pH 48 hours after inclusion | 48 hours after inclusion
  Hematosis
pH 72 hours after inclusion | 72 hours after inclusion
  Hematosis
pH 7 days after inclusion | 7 days after inclusion
  Hematosis
PaCO2 before each PP session | Up to Day 28
  Hematosis
PaCO2 1 hour after PP initiation at each PP session | Up to Day 28
  Hematosis
PaCO2 6 hours after PP initiation at each PP session | Up to Day 28
  Hematosis
PaCO2at the end of each PP session | Up to Day 28
  Hematosis
PaCO2 4 hours after return to supine after each PP session | Up to Day 28
  Hematosis
PaCO2 48 hours after inclusion | 48 hours after inclusion
  Hematosis
PaCO2 72 hours after inclusion | 72 hours after inclusion
  Hematosis
PaCO2 7 days after inclusion | 7 days after inclusion
  Hematosis
Plateau pressure (Pplat) before each PP session | Up to Day 28
  Protective mechanical ventilation
Plateau pressure (Pplat) 1 hour after PP initiation at each PP session | Up to Day 28
  Protective mechanical ventilation
Plateau pressure (Pplat) 6 hours after PP initiation at each PP session | Up to Day 28
  Protective mechanical ventilation
Plateau pressure (Pplat) at the end of each PP session | Up to Day 28
  Protective mechanical ventilation
Plateau pressure (Pplat) 4 hours after return to supine after each PP session | Up to Day 28
  Protective mechanical ventilation
Plateau pressure (Pplat) 48 hours after inclusion | 48 hours after inclusion
  Protective mechanical ventilation
Plateau pressure (Pplat) 72 hours after inclusion | 72 hours after inclusion
  Protective mechanical ventilation
Plateau pressure (Pplat) 7 days after inclusion | 7 days after inclusion
  Protective mechanical ventilation
Positive Expiratory Pressure (PEEP) before each PP session | Up to Day 28
  Protective mechanical ventilation
Positive Expiratory Pressure (PEEP) 1 hour after PP initiation at each PP session | Up to Day 28
  Protective mechanical ventilation
Positive Expiratory Pressure (PEEP) 6 hours after PP initiation at each PP session | Up to Day 28
  Protective mechanical ventilation
Positive Expiratory Pressure (PEEP) at the end of each PP session | Up to Day 28
  Protective mechanical ventilation
Positive Expiratory Pressure (PEEP) 4 hours after return to supine after each PP session | Up to Day 28
  Protective mechanical ventilation
Positive Expiratory Pressure (PEEP) 48 hours after inclusion | 48 hours after inclusion
  Protective mechanical ventilation
Positive Expiratory Pressure (PEEP) 72 hours after inclusion | 72 hours after inclusion
  Protective mechanical ventilation
Positive Expiratory Pressure (PEEP) 7 days after inclusion | 7 days after inclusion
  Protective mechanical ventilation
Driving Pressure (Δp) before each PP session | Up to Day 28
  Protective mechanical ventilation
Driving Pressure (Δp) 1 hour after PP initiation at each PP session | Up to Day 28,
  Protective mechanical ventilation
Driving Pressure (Δp) 6 hours after PP initiation at each PP session | Up to Day 28
  Protective mechanical ventilation
Driving Pressure (Δp) at the end of each PP session | Up to Day 28
  Protective mechanical ventilation
Driving Pressure (Δp) 4 hours after return to supine after each PP session | Up to Day 28
  Protective mechanical ventilation
Driving Pressure (Δp) 48 hours after inclusion | 48 hours after inclusion
  Protective mechanical ventilation
Driving Pressure (Δp) 72 hours after inclusion | 72 hours after inclusion
  Protective mechanical ventilation
Driving Pressure (Δp) 7 days after inclusion | 7 days after inclusion
  Protective mechanical ventilation
Tidal Volume (Vt) before each PP session | Up to Day 28
  Protective mechanical ventilation
Tidal Volume (Vt) 1 hour after PP initiation at each PP session | Up to Day 28
  Protective mechanical ventilation
Tidal Volume (Vt) 6 hours after PP initiation at each PP session | Up to Day 28
  Protective mechanical ventilation
Tidal Volume (Vt) at the end of each PP session | Up to Day 28
  Protective mechanical ventilation
Tidal Volume (Vt) 4 hours after return to supine after each PP session | Up to Day 28
  Protective mechanical ventilation
Tidal Volume (Vt) 48 hours after inclusion | 48 hours after inclusion
  Protective mechanical ventilation
Tidal Volume (Vt) 72 hours after inclusion | 72 hours after inclusion
  Protective mechanical ventilation
Tidal Volume (Vt) 7 days after inclusion | 7 days after inclusion
  Protective mechanical ventilation
Respiratory Rate (Fr) before each PP session | Up to Day 28
  Protective mechanical ventilation
Respiratory Rate (Fr) 1 hour after PP initiation at each PP session | Up to Day 28
  Protective mechanical ventilation
Respiratory Rate (Fr) 6 hours after PP initiation at each PP session | Up to Day 28
  Protective mechanical ventilation
Respiratory Rate (Fr) at the end of each PP session | Up to Day 28
  Protective mechanical ventilation
Respiratory Rate (Fr) 4 hours after return to supine after each PP session | Up to Day 28
  Protective mechanical ventilation
Respiratory Rate (Fr) 48 hours after inclusion | 48 hours after inclusion
  Protective mechanical ventilation
Respiratory Rate (Fr) 72 hours after inclusion | 72 hours after inclusion
  Protective mechanical ventilation
Respiratory Rate (Fr) 7 days after inclusion | 7 days after inclusion
  Protective mechanical ventilation
Esophageal pressure (for equipped sites) before each PP session | Up to Day 28
  Alveolar recruitment
Esophageal pressure (for equipped sites) 1 hour after PP initiation at each PP session | Up to Day 28
  Alveolar recruitment
Esophageal pressure (for equipped sites) at the end of each PP session | Up to Day 28
  Alveolar recruitment
Transpulmonary pressure (TPP) (for equipped sites) before each PP session | Up to Day 28
  Alveolar recruitment
Transpulmonary pressure (TPP) (for equipped sites) 1 hour after PP initiation at each PP session | Up to Day 28
  Alveolar recruitment
Transpulmonary pressure (TPP) (for equipped sites) at the end of each PP session | Up to Day 28
  Alveolar recruitment
Electrical Impedance Tomography data (for equipped sites) before each PP session | Up to Day 28
  Alveolar recruitment
Electrical Impedance Tomography data (for equipped sites) 1 hour after PP initiation at each PP session | Up to Day 28
  Alveolar recruitment
Electrical Impedance Tomography data (for equipped sites) at the end of each PP session | Up to Day 28
  Alveolar recruitment
Pneumothorax | Within the first 7 days
  Barotrauma
Pneumomediastinum | Within the first 7 days
  Barotrauma
Sub cutaneous emphysema | Within the first 7 days
  Barotrauma
Hospital mortality | At Day 28
Hospital mortality | At Day 90
Ventilator free days (VFD) | At Day 28
Ventilator free days (VFD) | At Day 90
Number of days alive without extra-respiratory organ failure | At Day 28
Number of days alive without extra-respiratory organ failure | At Day 90
Length of stay in intensive care unit | Maximum 3 months after inclusion (follow-up duration)
Length of hospital stay | Maximum 3 months after inclusion (follow-up duration)
Medical Research Council (MRC) | At day 28 or discharge

CONTACTS AND LOCATIONS:
Overall Officials: François Cremieux, Study Director — AP-HM
Locations (1):
- Service Médecine Intensive et Réanimation, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Papazian L, Aubron C, Brochard L, Chiche JD, Combes A, Dreyfuss D, Forel JM, Guerin C, Jaber S, Mekontso-Dessap A, Mercat A, Richard JC, Roux D, Vieillard-Baron A, Faure H. Formal guidelines: management of acute respiratory distress syndrome. Ann Intensive Care. 2019 Jun 13;9(1):69. doi: 10.1186/s13613-019-0540-9. PMID 31197492
- [Background] National Heart, Lung, and Blood Institute PETAL Clinical Trials Network; Moss M, Huang DT, Brower RG, Ferguson ND, Ginde AA, Gong MN, Grissom CK, Gundel S, Hayden D, Hite RD, Hou PC, Hough CL, Iwashyna TJ, Khan A, Liu KD, Talmor D, Thompson BT, Ulysse CA, Yealy DM, Angus DC. Early Neuromuscular Blockade in the Acute Respiratory Distress Syndrome. N Engl J Med. 2019 May 23;380(21):1997-2008. doi: 10.1056/NEJMoa1901686. Epub 2019 May 19. PMID 31112383
- [Background] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337